CLINICAL TRIAL: NCT01550237
Title: A Randomised, Two Centre Trial on Daily Cone-beam vs Standard Weekly Orthogonal Image Guided Radiotherapy (IGRT) for Prostate Cancer
Brief Title: Curative Image Guided Radiotherapy for Prostate Cancer
Acronym: RIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/710
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Prostatic Neoplasms
Keywords: radiotherapy, image-guided; adverse effects; position verification; safety margins
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiotherapy daily reduced (Experimental): radiotherapy, with daily CT position verification and reduced safety margins
  Interventions: Radiation: radiotherapy daily verification reduced safety margins
- radiotherapy weekly standard (Active Comparator): radiotherapy, with weekly orthogonal position verification and standard safety margins
  Interventions: Radiation: radiotherapy weekly verification standard safety margins

INTERVENTIONS:
Radiation: radiotherapy daily verification reduced safety margins — curative radiotherapy to 78 Gy in 39 fractions with daily CT position verification and reduced safety margins (7mm)
  Arms: radiotherapy daily reduced
Radiation: radiotherapy weekly verification standard safety margins — curative radiotherapy to 78 Gy in 39 fractions with weekly orthogonal position verification and standard safety margins (10-15 mm)
  Arms: radiotherapy weekly standard

SUMMARY:
The clinical importance of cone beam computer tomography based image guided radiotherapy (CT- IGRT) has not been established. The primary aim of the present trial is to investigate whether CT- IGRT and consequently reduced safety margins reduces the rectal side effects from curative, high dose radiotherapy in prostate cancer. Any impact of the reduced planning target volume in the CT- IGRT arm on biochemical freedom from disease will be evaluated as secondary outcome.

An open randomised phase III trial. The included men will be randomised to receive curative radiotherapy to 78 Gy in 39 fractions with weekly orthogonal position verification and standard safety margins (10-15 mm) or 78 Gy in 39 fractions with daily CT position verification and reduced safety margins (7mm).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed adenocarcinoma of prostate
* No evidence of nodal or distant metastases (N0M0)
* Intermediate or high risk based on T stage, PSA level and Gleason score
* Informed consent

Exclusion Criteria:

* Previous treatment for cancer last 5 years, except basal cell carcinoma of skin
* Any previous radiotherapy, except KV or electron treatment of skin tumors outside the pelvis
* Metallic hip joint replacement
* Pre-existing intestinal or genitourinary disease with increased risk of side effects
* Any pre-existing condition making the patient unsuitable for radiotherapy
* Any pre-existing condition making the patient unsuitable for hormonal therapy
* Any pre-existing condition making the patient unsuitable for MRI.
* ALAT, GT, ALP, creatinin > 1.5 x upper normal limit

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Acute rectal side effects | 10 weeks
  FWUO94

SECONDARY OUTCOMES:
Freedom from biochemical failure | 3 years
Overall survival | up to 10 years
Cancer specific survival | up to 10 years
Late genitourinary and rectal side effects | up to 10 years
Acute genitourinary side effects | 10 weeks
quality of life | up to 10 years
  HRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Jo Å Lund, MD PhD, Principal Investigator — St Olavs Hospital, University Hospital, Trondheim, Norway
Locations (2):
- Norway (2):
  - Ålesund Sykehus, Ålesund
  - St Olavs Hospital, Trondheim

REFERENCES:
- [Result] Tondel H, Lund JA, Lydersen S, Wanderas AD, Aksnessaether B, Jensen CA, Kaasa S, Solberg A. Radiotherapy for prostate cancer - Does daily image guidance with tighter margins improve patient reported outcomes compared to weekly orthogonal verified irradiation? Results from a randomized controlled trial. Radiother Oncol. 2018 Feb;126(2):229-235. doi: 10.1016/j.radonc.2017.10.029. Epub 2018 Feb 3. PMID 29398152